CLINICAL TRIAL: NCT04933032
Title: Prevalence and Risk Factors of Uterine Niche Following Different Caesarean Section Techniques:a Hospital Based Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Abdelrahman Faisal Abdellattif, Assistant lecturer of OB./GYN. sohag university hospitals, Sohag University
Other Study IDs: soh-med-21-04-17
Record Dates: First submitted 2021-06-13; First posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Appropriate Diagnostic Criteria of Uterine Niche With Detection of Prevalence , Risk Factors and Associated Symptomes
Keywords: niche , caesearan section scar defect , isthmocele

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this study is to institute clically relevant and objective sonographic criteria for the diagnosis of ceasearan section scar defect(CSSD) once the appropriate diagnostic criteria are established the natural history of CSSD could be elucidated through exploration of the prevelance ,risk factors, and associated symptomes of the disease

ELIGIBILITY:
Inclusion Criteria:

* all women underwent c-section

Exclusion Criteria:

* known uterine anomaly
* prior uterine surgery -prior uterine rupture
* chronic medical disease like diabetes -use of steroid over last year regularly
* obstetrical complications like multifetal pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All women undergoing a C-section will be asked to pariticpate in the study with follow up cases for 6 months
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
prevelance and risk factors of ceasearan section defects | one year
  follow up of women underwent their section for 6 monthes

CONTACTS AND LOCATIONS:
Locations (1):
- Abdelraman Fasial, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No